CLINICAL TRIAL: NCT00690989
Title: If You Build it, They Will Come; But Will They Return for Follow-up? A Retrospective Assessment of Potential Risk Factors for Patient Failure to Follow-up at a Community Based Headache Clinic
Brief Title: Retrospective Evaluation of Patient Failure to Follow-up at a Community Based Headache Clinic
Status: Completed | Type: Observational
Sponsor: Kilgo Headache Clinic (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Principal Investigator, Gary R. Kilgo, M. D., Medical director, Kilgo Headache Clinic
Other Study IDs: MK-0974 IISP #35151
Record Dates: First submitted 2008-06-03; First posted 2008-06-05 (Estimated); Last update posted 2015-04-03 (Estimated); Status verified 2015-03

CONDITIONS: Headache
Keywords: Headache; Adherence; Followup
MeSH Terms: conditions — Headache

STUDY DESIGN:
Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

SUMMARY:
This is a retrospective review of the records of patients seen at the Kilgo Headache Clinic in Alabama between 7/1/05 and 6/30/07. The goal of the study is to identify factors at the time of the initial office visit that can be used to predict failure to follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Headache
* Initial office visit between 7/1/05 and 6/30/07

Exclusion Criteria:

* None

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Community based headache clinic population
Sampling Method: Non-Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2005-07; Primary Completion 2007-06 (Actual); Study Completion 2009-06 (Actual)

PRIMARY OUTCOMES:
Adherence to followup recommendations | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Gary R. Kilgo, M.D., Principal Investigator — Kilgo Headache Clinic